CLINICAL TRIAL: NCT06620068
Title: Causal Association Between Plasma Vascular Endothelial Growth Factor Family Proteins and Placenta Previa: A Two-Sample Mendelian Randomization Study
Brief Title: Causal Relationship Between Plasma VEGF Family Proteins and Placenta Previa: A Two-Sample Mendelian Randomization Study
Acronym: VEGF PP
Status: Not yet recruiting | Type: Observational
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Collaborators: The Second People's Hospital of Foshan (Other); First People's Hospital of Foshan (Other); Maternal and Child Health Hospital of Foshan (Other)
Responsible Party: Principal Investigator, Zhibin Xu, Professor, Guangzhou Institute of Respiratory Disease
Other Study IDs: FSKY20240924
Record Dates: First submitted 2024-09-24; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Placenta Previa
Keywords: Vascular Endothelial Growth Factor (VEGF); Mendelian Randomization; Angiogenesis; Pregnancy Complications; Placental Development
MeSH Terms: conditions — Placenta Previa; Pregnancy Complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — The study utilizes genome-wide association study (GWAS) data from publicly available biobanks (e.g., UK Biobank and FinnGen), which include samples with DNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to investigate the causal relationship between plasma vascular endothelial growth factor (VEGF) family proteins and placenta previa using a two-sample Mendelian randomization (MR) approach. Genome-wide association study (GWAS) data will be analyzed to assess the correlation and potential causality between VEGF protein levels and the occurrence of placenta previa.

DETAILED DESCRIPTION:
Placenta previa is a serious complication during pregnancy, leading to significant risks for both the mother and the fetus. This study utilizes Mendelian randomization (MR) to explore the potential causal link between plasma levels of VEGF family proteins (including VEGFA, VEGFB, VEGFC, VEGFD, and PLGF) and the risk of placenta previa. By using genome-wide association study (GWAS) data from the UK Biobank and FinnGen datasets, the study aims to provide insights into the role of angiogenesis and abnormal placental development. The MR analysis will help minimize confounding factors and provide robust evidence regarding the causal relationship between VEGF proteins and placenta previa.

ELIGIBILITY:
Inclusion Criteria:

* Participants included in genome-wide association studies (GWAS) with available data on plasma VEGF family proteins and placenta previa.

Exclusion Criteria:

* Participants with incomplete or missing data on plasma VEGF levels or placenta previa.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study analyzes data from European populations included in genome-wide association studies (GWAS) from UK Biobank and FinnGen, focusing on individuals with available plasma VEGF family protein levels and placenta previa data.
Sampling Method: Non-Probability Sample
Enrollment: 207473 (Estimated)
Dates: Start 2024-09-25 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Causal relationship between plasma VEGFA levels and the risk of placenta previa | Data analysis and outcome assessment will be completed by December 2024
  This outcome measures the association between plasma VEGFA levels (measured in picograms per milliliter) and the occurrence of placenta previa, using Mendelian Randomization (MR) analysis to assess causality.

SECONDARY OUTCOMES:
Causal relationship between plasma VEGFB levels and the risk of placenta previa | Data analysis and outcome assessment will be completed by December 2024
  This outcome measures the association between plasma VEGFB levels (measured in picograms per milliliter) and the occurrence of placenta previa, using Mendelian Randomization (MR) analysis to assess causality.
Causal relationship between plasma VEGFC levels and the risk of placenta previa | Data analysis and outcome assessment will be completed by December 2024
  This outcome measures the association between plasma VEGFC levels (measured in picograms per milliliter) and the occurrence of placenta previa, using Mendelian Randomization (MR) analysis to assess causality.
Causal relationship between plasma PLGF levels and the risk of placenta previa | Data analysis and outcome assessment will be completed by December 2024
  This outcome measures the association between plasma PLGF levels (measured in picograms per milliliter) and the occurrence of placenta previa, using Mendelian Randomization (MR) analysis to assess causality.